CLINICAL TRIAL: NCT03790228
Title: Anlotinib Combined With Pemetrexed And Carboplatin Followed by Maintenance Therapy With Anlotinib Plus Pemetrexed as the First-line Treatment in Patients With Advanced Nonsquamous NSCLC
Brief Title: Anlotinib Combined With Pemetrexed And Carboplatin as First-line Treatment in Advanced Nonsquamous NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER L012
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2019-12

CONDITIONS: Non-squamous Cell Non-Small Cell Lung Cancer
Keywords: nonsquamous NSCLC; Anlotinib; Pemetrexed; Carboplatin; First-line
MeSH Terms: interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Intervention Model Description: Anlotinib combined with Pemetrexed and Carboplatin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Combined With Pemetrexed And Carboplatin (Experimental): Anlotinib(12mg, QD, PO, d1-14, 21 days per cycle) plus Pemetrexed (500mg/m2, IV, d15-21,21 days per cycle) and Carboplatin(AUC5,IV, d15-21,21 days per cycle,using 4 cycles)
  Interventions: Drug: Anlotinib Combined With Pemetrexed And Carboplatin

INTERVENTIONS:
Drug: Anlotinib Combined With Pemetrexed And Carboplatin — Anlotinib(12mg, QD, PO, d1-14, 21 days per cycle) plus Pemetrexed (500mg/m2, IV, d15-21,21 days per cycle) and Carboplatin(AUC5,IV, d15-21,21 days per cycle,using 4 cycles)

SUMMARY:
In recent years, with the progress in the treatment field, Non-Small Cell Lung Cancer(NSCLC) has become the most successful cancer species in precision medicine. Patients with positive driving genes such as EGFR, ALK, ROS1, BRAF and so on have clearly targeted drugs, which bring survival benefits to patients.However, about 50% of patients still lack a clear driving gene target, which has become the focus of current research.In the field of wild-type NSCLC with negative driver genes, the classic first-line treatment regimen is the two-drug regimen containing platinum.The study by Kimura T in the first-line treatment of 54 wild-type advanced NSCLC patients with carboplatin and pemetrexed showed that the ORR, mPFS and mOS of patients with wild-type non-squamous NSCLC treated with carboplatin permetrexine were 35.8%, 5.4 months and 12.7 months respectively.

Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development.In the phase Ⅲ study, patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib or placebo, the anlotinib group PFS and OS were 5.37 months and 9.46 months, the placebo group PFS and OS were 1.4 months and 6.37 months.

The efficacy and safety of Anlotinib combined with Pemetrexed and Carboplatin followed by maintenance therapy with Anlotinib plus Pemetrexed as the first-line treatment in patients with advanced nonsquamous NSCLC deserve further exploration.

DETAILED DESCRIPTION:
This is a multicentre single arm clinical trial conducted in China.The purpose of this study is to evaluate and observe Anlotinib (12mg,QD, PO d1-14, 21 days per cycle) combined with Pemetrexed(500mg/m2,IV,d15-21,21 days per cycle)and Carboplatin(AUC5,IV,d15-21,21 days per cycle,4 cycles) as the first-line treatment in patients with advanced nonsquamous NSCLC .After four cycles of induction,patients continued to receive Anlotinib and Pemetrexed.As the report,The median PFS of advanced NSCLC treated by Pemetrexed and Carboplatin was 6 months.We expect the median PFS of Anlotinib combined with Pemetrexed and Carboplatin as the first-line treatment in patients with advanced nonsquamous NSCLC was 10 months.Using PASS15, we calculated the sample size of this study was 34(α=0.05、β=0.2), according to 20% censoring,the expected sample size is 43.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form prior to patient entry;
* Male or female patients aged 18-75 years old;
* Diagnosed with advanced NSCLC (phase IIIB/IV) through pathology, Neoadjuvant chemotherapy, or postoperative adjuvant chemotherapy or neoadjuvant chemotherapy combined with postoperative adjuvant chemotherapy or targeted chemoradiotherapy for local advanced disease recurrence within 6 months after completion;
* In the past 3 months at least one target lesion that had not previously been irradiated,and at least one direction with the longest diameter at baseline greater than 10 mm (shorter diameter required not less than 15 mm if lymph nodes are involved)could be imaged by CT scan or MRI;
* Expected Survival Time: Over 6 months;
* Had an Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1 (on a 5-point scale, with higher scores indicating increasing disability);
* The main organs function are normally, the following criteria are met:(1)Blood routine examination criteria should be met (no blood transfusion and blood products within 14 days, no correction by G-CSF and other hematopoietic stimuli): HB≥90 g/L; ANC ≥ 1.5×10^9/L; PLT ≥80×10^9/L;(2)Biochemical examinations must meet the following criteria: TBIL<1.5×ULN; ALT and AST < 2.5×ULN, and for patients with liver metastases < 5×ULN; Serum Cr ≤ 1.25×ULN or endogenous creatinine clearance > 60 ml/min (Cockcroft-Gault formula);
* Women of child-bearing age should take appropriate contraceptive measures and should not breastfeed from screening to 3 months after stopping the study and treatment.Before starting administration, the pregnancy test was negative, or one of the following criteria was met to prove that there was no risk of pregnancy:

  1. Postmenopause is defined as amenorrhea at least 12 months after age 50 and cessation of all exogenous hormone replacement therapy;
  2. Postmenopausal women under the age of 50 May also be considered postmenopausal if their amenorrhea is 12 months or more after the cessation of all exogenous hormone therapy and their luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the reference value range of laboratory postmenopausal;
  3. Has undergone irreversible sterilization surgery, including hysterectomy, bilateral ovectomy or bilateral salpingectomy, except for bilateral tubal ligation.

For men, consent is required to use appropriate methods of contraception or to be surgically sterilized during the trial and 8 weeks after the last administration of the trial drug.

Exclusion Criteria:

* Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer),Lung sarcomatoid carcinoma;
* Had histologically confirmed lung squamous cell carcinoma, or adenosquamous carcinoma;
* Patients with pathological fracture in bone metastasis of non-small-cell lung cancer;
* Tumor histology or cytology confirmed EGFR mutagenesis [EGFR sensitive mutations include 18 exon point mutations (G719X), 19 exon deletions, 20 exon S768I mutations and 21 exon point mutations (L858R and L861Q)] and ALK gene rearrangement positivity, include EGFR/ALK status cannot be determined for various reasons;
* Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor;
* Medical history and combined history：

  1. Active brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 28 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms and metastases in midbrain, pons, cerebellum, medulla oblongata, or spinal cord, brain metastases and local radiotherapy after two weeks to allow group);
  2. The patient is participating in other clinical studies or completing the previous clinical study in less than 4 weeks;
  3. Had malignant tumors except NSCLC within 5 years before enrollment(except for patients with cervical carcinoma in situ , basal cell or squamous cell skin cancer who have undergone a curative treatment, local prostate cancer after radical resection, ductal carcinoma in situ or papillary thyroid cancer after radical resection);
  4. Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;Note: Under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose heparin (adult daily dose of 0.6 million to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg) is allowed for preventive purposes;
  5. Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
  6. The effects of surgery or trauma have been eliminated for less than 14 days before enrollment in subjects who have undergone major surgery or have severe trauma;
  7. Severe acute or chronic infections requiring systemic treatment;
  8. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
  9. There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma;
  10. Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment;
  11. Long-term unhealed wounds or fractures;
  12. Decompensated diabetes or other ailments treated with high doses of glucocorticoids;
  13. Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
  14. Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
  15. Events of venous/venous thrombosis occurring within the first 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* Physical examination and laboratory findings:

  1. A known history of HIV testing positive or acquired immunodeficiency syndrome (AIDS);
  2. Untreated active hepatitis (hepatitis b: HBsAg positive and HBV DNA more than 1 x 103 copy /ml; Hepatitis c: HCV RNA is positive and liver function is abnormal); Combined with hepatitis b and hepatitis c infection;
  3. Serious diseases that endanger patients' safety or affect patients' completion of research,according to the researchers' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival，PFS | each 42 days up to PD or death(up to 24 months)
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate,ORR | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate,DCR | each 42 days up to intolerance the toxicity or PD (up to 24 months).
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Overall Survival,OS | each 42 days up to intolerance the toxicity or PD (up to 24 months) .
  Defined as the time until death due to any cause.
Safety(Number of Participants with Adverse Events ) | each 42 days up to intolerance the toxicity or PD (up to 24 months).
  Number of Participants with Adverse Events.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China